CLINICAL TRIAL: NCT00212771
Title: Long-Term Efficacy and Safety Evaluation of Asenapine (10-20 mg/Day) in With Schizophrenia or Schizoaffective Disorder, in a Multicenter Trial Using (10-20 mg/Day) as a Control
Brief Title: Efficacy and Safety of Asenapine Using an Active Control in Subjects With Schizophrenia or Schizoaffective Disorder (25520)(P05846)
Acronym: ACTAMESA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05846; 25520
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: asenapine
- Arm 2 (Active Comparator)
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: asenapine — Flexible dose, 1-2 tablets sublingual two times per day (1 or 2 tablets in the morning and 1 or 2 tablets in the evening). Each tablet contains either 5 mg asenapine or matching placebo.
  Other Names: Org 5222; SCH 900274
  Arms: Arm 1
Drug: olanzapine — Flexible dose, 1-2 capsules oral once per day (in the morning). Each capsule contains 10 mg olanzapine or matching placebo.
  Other Names: Zyprexa
  Arms: Arm 2

SUMMARY:
The primary features of schizophrenia and schizoaffective disorder are positive (inability to think clearly and distinguish reality from fantasy) and negative symptoms (reduction or absence of normal behavior or emotions). Other symptoms include reduced ability to recall and learn information, difficulty in problem solving maintaining productive employment.

Asenapine is an investigational drug that may help to correct the above schizophrenia by altering the inbalance of brain hormones such as dopamine serotonin. This is a long-term extension trial to further test the efficacy and safety asenapine and a comparator agent (olanzapine) in the treatment of patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Subject with schizophrenia or schizoaffective disorder. Must have completed 12 months treatment under protocol 25517. Subject must sign a written informed consent.

Exclusion Criteria:

* Have an uncontrolled, unstable, clinically significant medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2004-09; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change in total PANSS score at endpoint | Screening, Week 76, 100, and once every 24 weeks thereafter until endpoint

SECONDARY OUTCOMES:
Changes in PANSS subscale scores and Marder factor scores | Every 24 weeks after baseline
Changes in CGI-S | Every 12 weeks after baseline
Patient functionality and subjective well-being (as measured by LOF, SF-12 and SWN) | Every 48 weeks after baseline
Severity of depressed mood (as measured by the Calgary Depression Scale for Schizophrenia) | Every 24 weeks after baseline
Resource utilization (as measured by frequency and length of hospital stay) | During the entire study period
Safety and tolerability: EPS (AIMS, BARS, SARS) | Every 24 weeks after baseline
Adverse Events | Continuously and up to 7 days after endpoint
Pregnancy Test | At endpoint
Blood Tests | Every 12 weeks after baseline
Weight and vital signs | Every 4 weeks after baseline
ECGs | Every 24 weeks after baseline

REFERENCES:
- [Result] Schoemaker J, Stet L, Vrijland P, Naber D, Panagides J, Emsley R. Long-term efficacy and safety of asenapine or olanzapine in patients with schizophrenia or schizoaffective disorder: an extension study. Pharmacopsychiatry. 2012 Jul;45(5):196-203. doi: 10.1055/s-0031-1301310. Epub 2012 Mar 27. PMID 22454251